CLINICAL TRIAL: NCT06167135
Title: Polycystic Ovary Syndrome, Insulin Resistance, Infertility, Obesity, and the Associated Mitochondrial Dysfunction With These Disorders in Hungarian Patients
Brief Title: Polycystic Ovary Syndrome, Mitochondrial Dysfunction, Obesity, Insulin Resistance Infertility (POMODORI) Cohort
Acronym: POMODORI
Status: Recruiting | Type: Observational
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Várbíró Szabolcs, University professor, Semmelweis University
Other Study IDs: 15672-6/2022/EÜIG
Record Dates: First submitted 2023-12-03; First posted 2023-12-12 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Infertility, Female; Polycystic Ovary Syndrome; Insulin Resistance; Primary Ovarian Insufficiency; Mitochondrial Alteration; Obesity
Keywords: Polycystic Ovary Syndrome; Insulin Resistance; Female Infertility; Obesity; Mitochondrial Dysfunction; Mitochondrial Alteration; Primary Ovarian Insufficiency
MeSH Terms: conditions — Infertility, Female; Polycystic Ovary Syndrome; Insulin Resistance; Primary Ovarian Insufficiency; Obesity; Mitochondrial Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Years
Biospecimen Retention: Samples With DNA — DNA isolated from blood sample and urine sample (urine epithelial cells)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Enrolling of 150 female patients of fertile age diagnosed with PCOS, insulin resistance, infertility, or mitochondrial disease, and the same number of age- and sex-matched controls are planned.

During the research biomarkers already with mitochondrial dysfunction in the scientific literature and common mtDNA abnormalities (deletions, point mutations, copy number changes, etc.) are examined.

DETAILED DESCRIPTION:
Mitochondrial dysfunction can be involved in the development of clinically heterogeneous diseases affecting multiple tissues and organs and can manifest at any age. Clinical signs are mainly manifested in the most energy-demanding tissues, such as the central nervous system, striated muscles, cardiac musculature, endocrine glands, liver, kidney, and sensory organs.

Polycystic ovarian syndrome (PCOS) is a multifactorial disorder with endocrine dysfunction characterized by ovulatory dysfunction, obesity, insulin resistance (IR), hirsutism, mild persistent inflammation, and ultrasonographically confirmed polycystic ovarian morphology. PCOS affects 5-15% of women of reproductive age. PCOS and IR are also common and treatable causes of infertility. As a result of delaying childbearing until later in life, this problem is affecting more and more couples. In the present study, the investigators hypothesize that PCOS, IR, and infertility associated with these conditions may also be a manifestation of mitochondrial dysfunction, the role of mitochondrial dysfunction in these conditions has been investigated to a limited extent based on the current literature.

Recent literature has shown that mitochondrial dynamics and morphology are two of the major factors in the development of insulin resistance and diabetes mellitus by regulating glucose metabolism. The investigators of this study cohort hypothesize that PCOS and IR may also be a manifestation of a primary mitochondrial pathology, the prevalence of IR and PCOS in primary mitochondrial patients has not yet been investigated based on the current literature. Recent literature suggests that mitochondrial dynamics and morphology are two of the main factors in the development of insulin resistance and diabetes mellitus by regulating glucose metabolism.

In the present experimental design, mitochondrial dynamics, bioenergetics, and autophagy pathways are hypothesized to play a key role in the pathomechanisms of PCOS and IR. A better understanding of the role of mitochondrial pathways in the pathophysiology of PCOS and IR may help to develop new biomarkers or therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

* Presence of polycystic ovary syndrome (PCOS) or insulin resistance (IR) associated with other multisystemic phenotypes, mitochondrial dysfunction
* history of infertility associated with other multisystemic phenotypes, mitochondrial dysfunction
* a known history of mitochondrial dysfunction and PCOS and/or IR
* general health is good and there is no serious general medical condition that would prevent participation would make participation highly risky

Exclusion Criteria:

* poor cooperation
* refusal to participate in the study

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Female patients of fertile age (between 20-45 years) who are being treated for insulin resistance and/or polycystic ovary syndrome, infertility, multi-organ symptoms, or possible primary ovarian insufficiency.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-09-10 (Actual); Primary Completion 2033-09-30 (Estimated); Study Completion 2033-09-30 (Estimated)

PRIMARY OUTCOMES:
Serum Glucose and Insulin Levels | One year
  The serum glucose and insulin levels are calculated by using plasma concentrations of insulin and glucose obtained during 120 min of a standard (75 g glucose) OGTT. Fasting, 1h and 2h glucose and insulin levels are measured
Clinical Pregnancy Rate | One year
  Clinical pregnancy rate = the number of clinical pregnancies/the total number of participants in the patient cohort × 100%

SECONDARY OUTCOMES:
Baseline Female Sex Hormone Levels and Thyroid Hormone Levels | One year
  Measurement of the baseline female sex hormone: anti-Mullerian hormone (AMH), luteinizing hormone (LH), follicle-stimulating hormone (FSH), estradiol, progesterone, total testosterone, free testosterone, SHBG) and thyroid hormone levels (thyroid stimulating hormone (TSH), T3, T4 + anti-thyroid peroxidase antibody, anti-thyroglobulin antibody) - in the unit of measurement used for the hormone concerned

OTHER OUTCOMES:
Body Mass Index (BMI) | One year
  The body mass index (BMI) is the metric currently in use for defining anthropometric height/weight characteristics in adults and classifying (categorizing) them into groups (expressed in kg/m2).
Metformin dose | One year
  Daily dose of metformin used (expressed in milligrams)
GLP-1 receptor agonist dose | One year
  Daily or weekly dose of the used glucagon-like peptide-1 (GLP-1) agonist depending on the exact type of active substance (expressed in milligrams)

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No